CLINICAL TRIAL: NCT01183845
Title: A Pilot Study to Evaluate the Applicability of the Crohn's Disease Endoscopy Index of Severity to Data Obtained by the Colonic Capsule Endoscopy in Ileocolonic Crohn's Disease
Brief Title: Evaluation of the Applicability of the CDEIS to Data Obtained by the Colonic Capsule Endoscopy in Crohn Disease
Acronym: CAPSCOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GETAID 2008-2
Record Dates: First submitted 2009-09-11; First posted 2010-08-18 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2011-08

CONDITIONS: Crohn Disease
Keywords: Crohn Disease; Crohn's Disease Endoscopy Index of Severity; Colon Capsule Endoscopy; Crohn's Disease located in colon and/or ileum
MeSH Terms: conditions — Crohn Disease | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exam with colon capsule (Experimental): Colon Capsule Endoscopy
  Interventions: Procedure: Colon Capsule Endoscopy

INTERVENTIONS:
Procedure: Colon Capsule Endoscopy — Ileocolonic endoscopy scheduled; then colon capsule endoscopy performed.

SUMMARY:
The Crohn's Disease Endoscopic Index of Severity is a validated index to assess the severity of ileocolonic lesions. Depth of ulcerations are evaluated in each segment of ileocolon and the surface of lesions and ulcerations are reported on a 10-cm analogic scale. The Crohn's Disease Endoscopic Index of Severity is the main score used in controlled trials to assess the endoscopic severity of lesions in Crohn's Disease.

The investigators aim to conduct a prospective pilot study primarily to evaluate the applicability of the Crohn's Disease Endoscopic Index of Severity to data obtained by the colonic capsule endoscopy procedure, provided that conventional ileo-colonoscopy and capsule endoscopy lead to comparable overall severity evaluations.

Secondary objectives are to assess reproducibility of the reading of data obtained by CCE and to compare these data with those obtained by conventional ileocolonoscopy. If overall severity evaluations derived from the two examinations are not comparable, the secondary objectives will be used in an attempt to understand the reasons of this discrepancy.

DETAILED DESCRIPTION:
Twenty-four patients with CD will be included in the study on the basis of the need for an ileo-colonoscopy whatever the indication.

* Males and females patients more than 18-years-old
* Known colonic CD patients with a diagnosis based on established clinical, endoscopic, ra-diologic, and histologic criteria
* Ileocolonoscopy scheduled
* Patients' agreement for the CCE procedure to be performed within the week following the ileocolonoscopy.
* Previous imaging of small bowel (one or more) by Small Bowel Follow Through (SBFT), Magnetic Resonance Enteroclysis (MRE) or Computed Tomography Enterography (CTE) performed in the last 12 months

ELIGIBILITY:
Inclusion Criteria:

* Males and females patients more than 18-years-old
* Known colonic CD patients with a diagnosis based on established clinical, endoscopic, ra-diologic, and histologic criteria
* Ileocolonoscopy scheduled
* Patients' agreement for the CCE procedure to be performed within the week following the ileocolonoscopy

Exclusion Criteria:

* Surgery of one or more segment of the colon or terminal ileum
* Non colonic CD
* High risk for capsule retention defined by the presence of clinically significant obstructive symptom related to intestinal or colonic stricture detected by small bowel imaging
* Stenosis of the colon or ileum not passed by the colonoscope
* Treatment with antiTNF or biotherapy after the ileocolonoscopy and before the CCE procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Data obtained by the colon capsule endoscopy as a Measure of safety | 1 month

SECONDARY OUTCOMES:
Reproducibility of the identification of the different anatomic segments on the CCE recordings | 1 month
Reproducibility of the detection of each lesion | At inclusion

CONTACTS AND LOCATIONS:
Overall Officials: LEMANN Marc, Study Director — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Alain ATTAR, MD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (3):
- France (3):
  - Hopital Beaujon, Clichy
  - Chru Lille, Lille
  - Chu Nantes, Nantes

REFERENCES:
- [Result] Casellas F, Vivancos JL, Sampedro M, Malagelada JR. Relevance of the phenotypic characteristics of Crohn's disease in patient perception of health-related quality of life. Am J Gastroenterol. 2005 Dec;100(12):2737-42. doi: 10.1111/j.1572-0241.2005.00360.x. PMID 16393228
- [Result] Itzkowitz SH, Harpaz N. Diagnosis and management of dysplasia in patients with inflammatory bowel diseases. Gastroenterology. 2004 May;126(6):1634-48. doi: 10.1053/j.gastro.2004.03.025. PMID 15168373
- [Result] Rutgeerts P, Diamond RH, Bala M, Olson A, Lichtenstein GR, Bao W, Patel K, Wolf DC, Safdi M, Colombel JF, Lashner B, Hanauer SB. Scheduled maintenance treatment with infliximab is superior to episodic treatment for the healing of mucosal ulceration associated with Crohn's disease. Gastrointest Endosc. 2006 Mar;63(3):433-42; quiz 464. doi: 10.1016/j.gie.2005.08.011. PMID 16500392
- [Result] Rutter M, Saunders B, Wilkinson K, Rumbles S, Schofield G, Kamm M, Williams C, Price A, Talbot I, Forbes A. Severity of inflammation is a risk factor for colorectal neoplasia in ulcerative colitis. Gastroenterology. 2004 Feb;126(2):451-9. doi: 10.1053/j.gastro.2003.11.010. PMID 14762782
- [Result] Triester SL, Leighton JA, Leontiadis GI, Fleischer DE, Hara AK, Heigh RI, Shiff AD, Sharma VK. A meta-analysis of the yield of capsule endoscopy compared to other diagnostic modalities in patients with obscure gastrointestinal bleeding. Am J Gastroenterol. 2005 Nov;100(11):2407-18. doi: 10.1111/j.1572-0241.2005.00274.x. PMID 16279893
- [Result] Kahn JL, Sick H, Laude M, Koritke JG. [Vascularization of the adipose body of the cheek]. Arch Anat Histol Embryol. 1990;73:3-20. French. PMID 1669678
- [Result] Eliakim R, Fireman Z, Gralnek IM, Yassin K, Waterman M, Kopelman Y, Lachter J, Koslowsky B, Adler SN. Evaluation of the PillCam Colon capsule in the detection of colonic pathology: results of the first multicenter, prospective, comparative study. Endoscopy. 2006 Oct;38(10):963-70. doi: 10.1055/s-2006-944832. PMID 17058158
- [Result] Schoofs N, Deviere J, Van Gossum A. PillCam colon capsule endoscopy compared with colonoscopy for colorectal tumor diagnosis: a prospective pilot study. Endoscopy. 2006 Oct;38(10):971-7. doi: 10.1055/s-2006-944835. PMID 17058159
- [Result] Mary JY, Modigliani R. Development and validation of an endoscopic index of the severity for Crohn's disease: a prospective multicentre study. Groupe d'Etudes Therapeutiques des Affections Inflammatoires du Tube Digestif (GETAID). Gut. 1989 Jul;30(7):983-9. doi: 10.1136/gut.30.7.983. PMID 2668130
- [Result] Modigliani R, Mary JY, Simon JF, Cortot A, Soule JC, Gendre JP, Rene E. Clinical, biological, and endoscopic picture of attacks of Crohn's disease. Evolution on prednisolone. Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives. Gastroenterology. 1990 Apr;98(4):811-8. doi: 10.1016/0016-5085(90)90002-i. PMID 2179031
- See also: Related Info — http://www.getaid.org